CLINICAL TRIAL: NCT03419039
Title: A Randomized, 24-week Parallel-group Placebo-controlled Multicenter (Phase 2) Study of Anthocyanins in People at Risk for Dementia
Brief Title: Anthocyanins as Dementia Prevention?
Acronym: ACID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SUSID656
Record Dates: First submitted 2018-01-15; First posted 2018-02-01 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-04

CONDITIONS: Dementia; Inflammation; Mild Cognitive Impairment; Coronary Artery Disease
Keywords: Mild Cognitive Impairment
MeSH Terms: conditions — Dementia; Inflammation; Cognitive Dysfunction; Coronary Artery Disease | interventions — Anthocyanins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anthocyanins (Experimental): Medox. 2 capsules x 2 daily, 320 mg daily.
  Interventions: Dietary Supplement: Anthocyanins
- Placebo (Placebo Comparator): 2 identically appearing placebo capsules daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Anthocyanins — Medox tablet containing 80 mg anthocyanins.
  Other Names: Medox 80 mg
  Arms: Anthocyanins
Dietary Supplement: Placebo — Identically appearing capsules.
  Arms: Placebo

SUMMARY:
The aim of this project is to study the safety and efficacy of anthocyanins in improving key dementia-related mechanisms and cognitive functioning in older people at risk for dementia. Secondary analyses will include a variety of biological measures, including biochemistry, imaging and cardiovascular measures.

DETAILED DESCRIPTION:
Design, Method, Material. Design: This is a randomized, 6-month, placebo-controlled Phase 2 study of anthocyanins (Medox) in people with increased risk for dementia, to explore the effects of anthocyanins on cognitive performance and a range of biological markers including blood markers of inflammation and oxidative stress, antioxidants, lipid profile, urine, faeces, and cardiovascular functions.

Method: Patients will be randomized (by means of a computerized program) to identically appearing capsules with Medox or placebo, 1:1 (produced by MedPalett). Patients will undergo monthly cognitive testing online. Brain MRI, structural and functional, will be performed before study start and at week 24. FDG-PET will also be done at sudy-start and study-end in a sub-group. Blood samples for analyses will be drawn at study start, after 12 weeks and at study end (week 24). Lumbar puncture for cerebrospinal fluid (CSF) analyses, and faeces analyses and urine will be done at study-start and study end, and additionally at week 12 for feces and urine. Cardiovascular test inlude cardio ankle vascular index (CAVI), and photopletysmography (PPG) measurements will be done at study start (baseline) week 2, 6, 12 and at study end (week 24). In a sub-group Flow mediated dilatation of brachial artery (FMD) will be done at study start, week 12 and study end.

The cognitive assessment battery consists of the CogTrack, an online cognitive test battery with proven utility, reliability, sensitivity and validity and sensitivity to change. The battery consists of ten subtests, which, based on factor analysis, are combined into the following domains: attention, memory and cognitive speed. The 15 word lists of the verbal memory test have been translated into Norwegian. The primary outcome measure will be the Quality of Episodic Memory combination of 2 accuracy scores from each of immediate and delayed word recall, word and picture recognition (4 tasks in total), which has been shown to be sensitive to cognitive changes . The battery will be administered online monthly at home, or with assistance from a research associate at SESAM/local research site if Internet is not available at home. Collection and registration will be performed securely online.

Patients will be tested at the same time of day on all occasions, usually in the morning. Testing procedures will be standardized (i.e. temperature, room, research associate, coffee intake).

Protocol amendment 17.08.20 Study: A randomized, 24-week parallel-group placebo-controlled multicenter (Phase 2) study of anthocyanins in people at risk for dementia.

Background for amendment Due to the COVID-19 pandemic, which has led to disease and even death within the Wesnes Cognition Ltd and contracted developers supporting the CogTrack cognitive testing, the maintenance of the CogTrack platform suffered and went fully down in June 2020. Accordingly participants were unable to access the platform and unable to complete the cognitive testing as part of the ACID study. A lot of resources were directed towards correcting the challenges. We have now been able to set up a different but nearly identical system, eCogPro, as an alternative test system. This system is expected to be ready to be administered to the participants in late August or early September.

Because of this inclusion of new participants has stopped, after having randomized 206 participants. There are 27 ongoing participants who have scheduled cognitive testing from today and until early October. The company producing active and placebo capsules, MedPalett, has agreed to distribute additional capsules to the remaining participants, enabling them to continue treatment until the cognitive test platform is up and running. Staff at MedPalett are unblended to allocation, and based on the study ID list of the remaining participants, will be able to deliver the correct capsules to study participants.

Other assessments, including physical testing and biomarker collection, are now running as normal, after having been shut down during the midst of the pandemic in April and May.

There have not been any safety concerns in the study so far, and no additional safety procedures will be initiated.

Amendment summary:

Participants who are still in the study will continue treatment up to 4 weeks beyond the scheduled 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* On none, or stable medication for the past three months AND
* Mild cognitive impairment (MCI) according to Winblad OR
* having >2 of the following conditions known to be associated with increased risk of cognitive impairment and dementia:
* stable cardiovascular disease defined as coronary artery disease (CAD) seen on angiogram
* cerebrovascular disease according to MRI criteria (i.e. presence of: Fazekas score >2 points OR cerebral infarct (>1 lesion) OR lacunar infarct (>1 lesion) OR lobar microbleed (>1 lesion), as judged by a qualified neuroradiologist) OR as visualized on CT scan for those having contraindications to MRI.
* hypercholesterolemia/significant cardiovascular risk, operationalized as use of statin at baseline
* hypertension, operationalized as previous diagnosis of arterial hypertension and/or use of antihypertensive drugs
* diabetes mellitus type 1
* metabolic syndrome including overweight (BMI>25) and diabetes mellitus type 2 (i.e. history of - and/or use of oral antidiabetic drugs and/or HbA1c >6.5%)

Exclusion Criteria:

* Any dementia (defined as CDR >0.5)
* Other known relevant brain disease such as Parkinson's disease, normal pressure hydrocephalus and other diseases which according to the study physician may cause cognitive decline
* Clinically significant depression, i.e. major depression or GDS-15 score > 7
* Unstable coronary heart disease
* Heart failure in need of treatment
* Systemic inflammatory diseases
* Other serious disease with expected survival <5 years
* Somatic disease that might affect cognitive function adversely
* Usage of heparin, warfarin and Non-Vitamin K Antagonist Oral Anticoagulants (NOAC)
* Any use of Medox during the 12 months prior to inclusion

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Quality of episodic memory. | Baseline to 24 weeks
  A composite measure from the CogTrack battery

SECONDARY OUTCOMES:
Secondary endpoints from CogTrack | Baseline to 24 weeks
  CogTrack evaluates attentional intensity index, sustained intensity index, cognitive reaction time, attentional fluctuation index, quality of working memory, quality of episodic memory and speed of memory retrieval.
Blood outcome analysis | Baseline to 24 weeks
  Lipid profile, fatty acids, cytokines ( among others: IL-1, IL-2, IL-6, TNF-a), plasma antoxidant status and vitamins (lipid peroxidation markers, vitamins E, C, A, total plasma antioxidant capacity, glutathion)., carinthine, blood glucose, HbA1c, anthocyanins and metabolites, mapping of a-beta degradation products.
Cardiovascular parameters | Baseline to 24 weeks
  Flow-mediated dilation (FMD), Cardiac-ankle vascular index (CAVI), photoplethysmogram (PPG).
Fecal analysis | Baseline to 24 weeks
  Microbiota
Urine analysis | Baseline to 24 weeks
  kyrinin
CSF measurements | Baseline to 24 weeks
  anthocyanin metabolites
MR-imaging/CT | Baseline to 24 weeks
  Diagnosing and follow-up of cerebrovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Dag Aarsland, MD., PhD., Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Lucia C, Tovar-Rios DA, Khalifa K, Kvernberg SM, Pola I, Bergland AK, Maple-Grodem J, Siow R, Ashton N, Ballard C, Thuret S, Aarsland D. Effects of Oral Anthocyanin Supplementation on In Vitro Neurogenesis, Hippocampus-Dependent Cognition, and Blood-Based Dementia Biomarkers: Results from a 24-Week Randomized Controlled Trial in Older Adults At Risk for Dementia (ACID). Nutrients. 2025 Aug 19;17(16):2680. doi: 10.3390/nu17162680. PMID 40871708
- [Derived] Borda MG, Ramirez-Velez R, Botero-Rodriguez F, Patricio-Baldera J, de Lucia C, Pola I, Barreto GE, Khalifa K, Bergland AK, Kivipelto M, Cederholm T, Zetterberg H, Ashton NJ, Ballard C, Siow R, Aarsland D; NJ FINGER. Anthocyanin supplementation in adults at risk for dementia: a randomized controlled trial on its cardiometabolic and anti-inflammatory biomarker effects. Geroscience. 2025 May 2. doi: 10.1007/s11357-025-01669-8. Online ahead of print. PMID 40314845
- [Derived] Aarsland D, Khalifa K, Bergland AK, Soennesyn H, Oppedal K, Holteng LBA, Oesterhus R, Nakling A, Jarholm JA, de Lucia C, Fladby T, Brooker H, Dalen I, Ballard C. A Randomised Placebo-Controlled Study of Purified Anthocyanins on Cognition in Individuals at Increased Risk for Dementia. Am J Geriatr Psychiatry. 2023 Feb;31(2):141-151. doi: 10.1016/j.jagp.2022.10.002. Epub 2022 Oct 18. PMID 36372613
- [Derived] Khalifa K, Bergland AK, Soennesyn H, Oppedal K, Oesterhus R, Dalen I, Larsen AI, Fladby T, Brooker H, Wesnes KA, Ballard C, Aarsland D. Effects of Purified Anthocyanins in People at Risk for Dementia: Study Protocol for a Phase II Randomized Controlled Trial. Front Neurol. 2020 Sep 2;11:916. doi: 10.3389/fneur.2020.00916. eCollection 2020. PMID 32982933